CLINICAL TRIAL: NCT02663869
Title: Aging With HIV at Younger vs Older Age: a Diverse Population With Distinct Comorbidity Profiles
Acronym: Aging_in_HIV
Status: Completed | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Giovanni Guaraldi, MD, University of Modena and Reggio Emilia
Other Study IDs: Aging with HIV
Record Dates: First submitted 2015-12-21; First posted 2016-01-26 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: HIV Infection; Aging
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV Aging-Young: 200 patients
- HIV Aging-Old: 200 patients
- controls: 1200 patients

SUMMARY:
Clinical hypotheses:

The increasing number of people aging with HIV is a matter of fact. Differences in prevalence of comorbidities between the general population and HIV-positive patients are mainly driven by duration of HIV infection rather than chronological age of HIV+ patients.

People aging with HIV display heterogeneous health conditions. Host factors and duration of HIV infection are associated with increased risk of MM, independently from chronological age and these factors are responsible of the prevalence difference of comorbidities and MM in comparison to the general population.

Objectives:

The study objective is to assess the prevalence of, and risk factors for, individual co-morbidities and multi morbidity (MM) between HIV-positive patients with similar duration of HIV infection, but 30 years difference. We compared estimates across both groups to a matched community-based cohort sampled from the general population.

DETAILED DESCRIPTION:
This study is a case-control study, including antiretroviral therapy (ART)-experienced patients, coming from the two following cohorts:

* Modena HIV Metabolic Clinic (MHMC) cohort and
* Romanian HIV cohort (RHC). For this study only patients living with HIV ≥ 20 years will belong to these two cohort. The Aging-Young patients acquired HIV infection in childhood, and Aging-old patients acquired HIV infection above the age of 30.

Aging-Young patients will be matched to Aging-Old patients considering gender and HIV duration (within 1 year interval) (This is the most important matching criteria. The exact number of year of HIV duration since HIV test is the major criteria). An HIV negative test within 5 years prior HIV diagnosis is required in the selection of patients from MHMC to avoid an unpredicted HIV time exposure in these patients.

Then, Aging-young and Aging-old patients will be age, gender matched with a 1: 3 ratio with CINECA (Consorzio Interuniversitario di Calcolo) "ARNO" records (control group, called "HIV-negative group"). The study will analyse 200 HIV Aging-Young and 200 HIV Aging-Old patients in comparison to 1200 controls.

In the first set of analyses, the prevalence of non-infectious comorbidities (NICM) and multimorbidities (MM) in HIV Aging-Young and in HIV Aging-Old groups will be compared to those of HIV-negative group using multivariable logistic regression models. In the second set of analyses, the probability of MM in the HIV Aging-Young cohort will be compared to the HIV Aging-Old one, using multivariable logistic regression models.

ELIGIBILITY:
Inclusion Criteria:

* HIV Aging-Old patients will be selected at Modena HIV metabolic Clinic. 200 consecutive patients who satisfy the following criteria:

  * HIV + since 20 year
  * HIV diagnosis occurred when the patient was older than 30 years
  * HIV negative test within 5 years prior HIV diagnosis
  * Multidisciplinary evaluation for comorbidities was performed during 2014
  * On HAART for at least 1 year
* HIV Aging-Young patients will be selected at Romanian HIV Cohort. 200 consecutive patients who satisfy the following criteria:

  * HIV + since 20 year
  * HIV diagnosis occurred when the patient was younger than 5 years
  * Multidisciplinary evaluation for comorbidities was performed during 2014
  * On HAART for at least 1 year

Exclusion Criteria:

* Not Applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV infected and not infected people
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Assess the prevalence of co-morbidities and multimorbidity between HIV-positive patients with similar duration of HIV infection, but 30 years difference | 1 year
  Multimorbidity is assessed by physician based on the concurrent presence of > 2 non infectious comorbidities (hypertension, cardiovascular disease, diabetes, etc)

CONTACTS AND LOCATIONS:
Locations (3):
- Department of Clinical Research of Holdsworth House Medical Practice, Sydney, Australia
- Univeristy of Modena and ReggioEmilia, Modena, Italy
- Hospital Clínic Per A La Recerca Biomèdica, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No